CLINICAL TRIAL: NCT04681404
Title: Assessment of Balance, Function and Quality of Life in Patients Before and After Knee Replacement
Brief Title: Balance After Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johannes Kepler University of Linz (Other)
Collaborators: Kepler University Hospital (Other)
Responsible Party: Principal Investigator, Christian Mittermaier, Christian Mittermaier, MD, Johannes Kepler University of Linz
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PMR_Knee TKA 001
Record Dates: First submitted 2020-02-12; First posted 2020-12-23 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Postural Balance; Knee Arthroplasty; Quality of Life
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Total Knee Arthroplasty (TKA) (Active Comparator): Patients intended to undergo surgery for total knee arthroplasty
  Interventions: Procedure: Knee Arthroplasty
- Unicompartmental Knee Arthroplasty (UKA) (Active Comparator): Patients intended to undergo surgery for unicompartmental knee arthroplasty
  Interventions: Procedure: Knee Arthroplasty
- Healthy Control (No Intervention)

INTERVENTIONS:
Procedure: Knee Arthroplasty — Comparison of TKA, UKA and healthy controls in relation to balance, function and QOL
  Arms: Total Knee Arthroplasty (TKA); Unicompartmental Knee Arthroplasty (UKA)

SUMMARY:
Evaluation of patients before and after knee arthroplasty regarding balance, function and quality of life. Comparison of total and unicompartmental knee arthroplasty. Comparison of the primary outcome parameter and selected secondary outcome parameters to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Primary gonarthrosis
* planned TKA or UKA
* adequate cognitive and lingual competence
* informed consent

Exclusion Criteria:

* TKA or UKA revision
* Surgery after trauma
* Rheumatic disease
* Neurologic disease
* previous arthroplasty of the lower extremity (<9 months)
* cardiovascular disease
* restricted weight bearing of the lower extremity after surgery

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Center of pressure track (COPT) | Before surgery
  Posturographic Parameter
Center of pressure track (COPT) | Day 3-7 after surgery
  Posturographic Parameter
Center of pressure track (COPT) | 3 months after surgery
  Posturographic Parameter
Center of pressure track (COPT) | 1 year after surgery
  Posturographic Parameter

SECONDARY OUTCOMES:
Functional reach test | Before surgery; day 3-7 after surgery; 3 months and 1 year after surgery
Timed up and go - test | Before surgery; day 3-7 after surgery; 3 months and 1 year after surgery
Knee Injury and Osteoarthritis Outcome Score | Before surgery; day 3-7 after surgery; 3 months and 1 year after surgery
  Scale: Points, Minimum: 0, Maximum: 100, higher score means better outcome
EQ-5D - Score | Before surgery; 1 year after surgery
  Scale: Points, Minimum: 1, Maximum: <0, higher score means better outcome
10 m Walking test | Before surgery; day 3-7 after surgery; 3 months and 1 year after surgery
WOMAC Score | Before surgery; 1 year after surgery, higher score means better outcome
  Scale: Points, Minimum: 0, Maximum: 240, higher score means worse outcome
Forgotten Joint Score | Before surgery; 1 year after surgery
  Scale: Points, Minimum: 0, Maximum: 100, higher score means better outcome
Oxford Knee Score | Before surgery; 1 year after surgery
  Scale: Points, Minimum: 12, Maximum: 60, higher score means worse outcome
Knee Society Score | Before surgery; 1 year after surgery
  Scale: Points, Minimum: 0, Maximum: 100, higher score means better outcome
The University of California at Los Angeles Activity Score | Before surgery; 1 year after surgery
  Scale: Points, Minimum: 1, Maximum: 10, higher score means better outcome
Area of Sway | Before surgery; day 3-7 after surgery; 3 months and 1 year after surgery
  Posturographic Parameter
Frequency of Sway | Before surgery; day 3-7 after surgery; 3 months and 1 year after surgery
  Posturographic Parameter
Harmony Index | Before surgery; day 3-7 after surgery; 3 months and 1 year after surgery
  Posturographic Parameter
Stability energy | Before surgery; day 3-7 after surgery; 3 months and 1 year after surgery
  Posturographic Parameter
Movement control | Before surgery; day 3-7 after surgery; 3 months and 1 year after surgery
  Posturographic Parameter
Feedback (visual, somatosensoric, vestibular) | Before surgery; day 3-7 after surgery; 3 months and 1 year after surgery
  Posturographic Parameter
Weight Distribution Index | Before surgery; day 3-7 after surgery; 3 months and 1 year after surgery
  Posturographic Parameter
Fulfillment of Tests | Before surgery; day 3-7 after surgery; 3 months and 1 year after surgery
  Posturographic Parameter

CONTACTS AND LOCATIONS:
Overall Officials: Christian Mittermaier, Dr, Principal Investigator — Kepler University Hospital
Locations (1):
- Kepler University Hospital, Linz, Austria